CLINICAL TRIAL: NCT04557150
Title: An Open-Label, Multicenter, Phase I Study Evaluating the Safety and Pharmacokinetics of Escalating Doses of Forimtamig (RO7425781) in Participants With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study Evaluating the Safety and Pharmacokinetics of Escalating Doses of Forimtamig in Participants With Relapsed or Refractory Multiple Myeloma (r/r MM)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BP42233; 2020-002012-46 (EudraCT Number); 2023-504571-25-00 (EU CTIS Number)
Record Dates: First submitted 2020-09-17; First posted 2020-09-21 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part I: Dose Escalation (Experimental): Participants will receive forimtamig as intravenous (IV) infusion and/or subcutaneous (SC) injection in a step-up dosing fashion.
  Interventions: Drug: Forimtamig
- Part II: Dose Expansion (Experimental): Dose Expansion cohorts with IV and/or SC administration, respectively, will be initiated at the Recommended Phase 2 Doses (RP2Ds) determined in Part I: Dose Escalation phase.
  Interventions: Drug: Forimtamig

INTERVENTIONS:
Drug: Forimtamig — Forimtamig will be administered via IV/SC administration. The RP2Ds determined during Part I: Dose Escalation will be administered during Part II: Dose Expansion. Forimtamig will be administered as per the dosing schedule defined in Part I.
  Other Names: RO7425781

SUMMARY:
This is a first-in-human, open-label, uncontrolled, multi-center, monotherapy, dose-escalation and dose expansion study. Forimtamig will be administered to participants with r/r MM for whom no standard-of-care treatment exists or who are intolerant to those established therapies. The study consists of two parts: dose-escalation of forimtamig (Part 1) and a randomized dose expansion of forimtamig (Part 2).

ELIGIBILITY:
Inclusion Criteria:

* Previously diagnosed with Multiple Myeloma (MM) based on standard criteria.
* Dose Escalation Phase and Dose Expansion Phase: Participants with r/r MM who have previously received therapy with an Immunomodulatory drug (IMiD) and Proteasome Inhibitor (PI) and are intolerant to or have no other option for standard-of-care treatment according to the Investigator.
* Life expectancy of at least 12 weeks.
* Agreement to provide protocol-specific biopsy material.
* AEs from prior anti-cancer therapy resolved to Grade =<1.
* Measurable disease.
* For female participants of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse), use contraceptive measures and refrain from donating eggs.
* For male participants: agreement to remain abstinent (refrain from heterosexual intercourse), use contraceptive measures and refrain from donating sperm.

Exclusion Criteria:

* Inability to comply with protocol-mandated hospitalization and activities restrictions.
* Pregnant or breastfeeding or intending to become pregnant during the study or within 3 months after last dose of study drug.
* Prior use of any monoclonal antibody, radioimmunoconjugate, or antibody-drug conjugate for MM treatment within 2 weeks before first forimtamig administration.
* Prior treatment with systemic immunotherapeutic agents within 2 weeks before first forimtamig administration.
* Treatment-related, immune-mediated AEs associated with prior immunotherapeutic agents.
* Treatment with radiotherapy, any chemotherapeutic agent, or treatment with any other anti-cancer agent (investigational or otherwise) within 2 weeks, prior to first forimtamig administration. Limited field palliative radiotherapy for bone pain or for soft tissue lesions is allowed.
* Autologous or allogeneic stem cell transplantation (SCT) within 100 days prior to first forimtamig infusion and/or signs of chronic graft versus host disease or ongoing immunosuppressive medication.
* Prior solid organ transplantation.
* Active auto-immune disease or flare within 6 months prior to start of study treatment
* Any medical condition or abnormality in clinical laboratory tests that, in the Investigator's or Medical Monitor's judgment, precludes the participant's safe participation in and completion of the study, or which could affect compliance with the protocol or interpretation of results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events (AEs) | Up to 104 weeks
Percentage of Participants with Dose Limiting Toxicities (DLTs) | Cycle 1 Day 1 up to Cycle 1 Day 35

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 104 weeks
Duration of Response (DOR) | Up to 104 weeks
Progression-Free Survival (PFS) | Up to 104 weeks
Overall Survival (OS) | Up to 104 weeks
Percentage of Participants with Anti-Drug Antibodies (ADAs) to Forimtamig | Up to 104 weeks
Maximum Concentration (Cmax) of Forimtamig | Up to 104 weeks
Time of Maximum Concentration (Tmax) of Forimtamig | Up to 104 weeks
Minimum Concentration (Cmin) of Forimtamig | Up to 104 weeks
SC Bioavailability (F) of Forimtamig | Up to 104 weeks
Apparent Clearance (CL/F) of Forimtamig | Up to 104 weeks
Volume of Distribution at Steady State (Vss) of Forimtamig (IV only) | Up to 104 weeks
Area Under the Curve (AUC) at Various Time Intervals of Forimtamig | Up to 104 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (20):
- Peter MacCallum Cancer Center, Melbourne, Victoria, Australia
- UZ Gent, Ghent, Belgium
- Denmark (2):
  - Rigshospitalet, København Ø
  - Odense Universitetshospital, Odense C
- France (3):
  - CHRU Lille - Hôpital Claude Huriez, Lille
  - CHU NANTES - Hôtel Dieu, Nantes
  - Hopital De Haut Leveque, Pessac
- Italy (4):
  - IRCCS Istituto Nazionale dei Tumori di Napoli - Pascale Ematologia Oncologica, Napoli, Campania
  - Policlinico S.Orsola-Malpighi, Bologna, Emilia-Romagna
  - Fond. IRCCS Istituto Nazionale Tumori, Milan, Lombardy
  - Instituto Clinico Humanitas, Rozzano, Lombardy
- New Zealand Clinical Research - Auckland, Auckland, New Zealand
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul St Mary's Hospital, Seoul
- Spain (3):
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Hospital Clinico Universitario de Salamanca, Salamanca
- United Kingdom (2):
  - St James University Hospital, Leeds
  - University College London Hospitals NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Eckmann J, Fauti T, Biehl M, Zabaleta A, Blanco L, Lelios I, Gottwald S, Rae R, Lechner S, Bayer C, Dekempe Q, Osl F, Carrie N, Kassem S, Lorenz S, Christopeit T, Carpy A, Bujotzek A, Broske AM, Dekhtiarenko I, Attig J, Kunz L, Cremasco F, Adelfio R, Fertig G, Dengl S, Gassner C, Bormann F, Kirstenpfad C, Kraft T, Diggelmann S, Knobloch M, Hage C, Feddersen R, Heidkamp G, Poschinger T, Mayoux M, Bernasconi L, Prosper F, Dumontet C, Martinet L, Leclair S, Xu W, Paiva B, Klein C, Umana P. Forimtamig, a novel GPRC5D-targeting T-cell bispecific antibody with a 2+1 format, for the treatment of multiple myeloma. Blood. 2025 Jan 9;145(2):202-219. doi: 10.1182/blood.2024025987. PMID 39476124